CLINICAL TRIAL: NCT06609980
Title: Fecal Microbiota Transplantation (Autologous) in Infants Treated with Antibiotics
Brief Title: Restoration of Antibiotics Related Infant Microbiota Perturbations by Autologous Fecal Transplant
Acronym: aFMT-babies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Maria Gloria Dominguez-Bello, Ph.D, Distinguished Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro2022001766
Record Dates: First submitted 2024-08-07; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Antibiotic Treatment
Keywords: FMT; autologous; children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Analysis will be done on de-identified samples so the outcomes assessor will be unaware
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Caregivers of the participants in the intervention arm will collect monthly fecal samples while the child is healthy and right before an antibiotic treatment which has been prescribed by the pediatrician for a non-gastrointestinal condition. One day after the last dose of antibiotics, the caregiver will collect another fecal sample and then the child will orally drink 2 ounces of the autologous fecal matter transplant inoculum prepared by the research team by mixing the child's own most recent sample prior to falling ill and mixed with milk. The caregivers then continue collecting samples once a week for a month followed by once a month for five months.
  Interventions: Drug: autologous fecal matter transplant
- Control (No Intervention): Participants do not partake in the autologous fecal matter transplant that will be used to re-seed the child's gut with his or her own personalized microbiome composition which was preserved prior to antibiotics use.

INTERVENTIONS:
Drug: autologous fecal matter transplant — Autologous fecal matter transplant will be used to re-seed the child's gut with his or her own personalized microbiome composition which was preserved prior to antibiotics use.
  Arms: Intervention Arm

SUMMARY:
Antibiotics are lifesaving therapeutic drugs which have been used by adults, children, and infants alike for decades. There is an increase in global use of antibiotics over the course of lifetime and earlier in lifetime, with some countries recording as high as 12 courses a year in children younger than two. While antibiotics are successful in eradicating many pathogenic bacteria, research has demonstrated significant effect on beneficial gut microbiota, including long-lasting shift in the dynamics, composition, richness, and maturity of the intestinal flora. Microbiota alterations during early life, including through antibiotics use as well as birth via C-section, constitute a developmental perturbation, which increases the risk of modern diseases of immune and metabolic dysfunction. Strong epidemiological evidence suggests associations between early stressors of the microbiota and a number of common diseases, such as obesity, asthma, allergies, celiac disease, and Type 1 Diabetes. Furthermore, excess antibiotic exposure is associated with the development of neurological and psychiatric disorders. Currently, no strategies exist to restore the microbiome other than reliance on spontaneous repair mechanism, which often takes months in a healthy individual barring further antibiotic exposure. Contrary to popular belief, ingestion of probiotics, particularly after antibiotics, has been demonstrated to slow down the repair as it introduces an exogenous and massive amounts of only a few types of bacterial strains into a finely-tuned ecosystem of hundreds of different strains.

It is hypothesized that by preserving the child's microbiome prior to antibiotic therapy and reintroducing it afterwards through an autologous fecal matter transplant (FMT) will assist in a quick, effective, and host-specific microbiome recolonization to the levels and patterns to those prior to antibiotics. This would in turn reduce the overall loss of microbiome diversity over the child's lifespan, essentially providing a 'reset' option to the child's most unadulterated version of microbiome. This approach utilizes delivering the sample by mixing it in maternal milk or formula and feeding it to the child through a bottle, which can be performed anywhere without any discomfort for the child.

DETAILED DESCRIPTION:
Antibiotics are lifesaving therapeutic drugs which have been used by adults, children, and infants alike for decades. There is an increase in global use of antibiotics over the course of lifetime and earlier in lifetime, with some countries recording as high as 12 courses a year in children younger than two. While antibiotics are successful in eradicating many pathogenic bacteria, research has demonstrated significant effect on beneficial gut microbiota, including long-lasting shift in the dynamics, composition, richness, and maturity of the intestinal flora.

Microbiota alterations during early life, including through antibiotics use as well as birth via C-section, constitute a developmental perturbation, which increases the risk of modern diseases of immune and metabolic dysfunction. Strong epidemiological evidence suggests associations between early stressors of the microbiota and a number of common diseases, such as obesity, asthma, allergies, celiac disease, and Type 1 Diabetes. There is evidence from mouse experiments of early perturbations in microbiota transmission at birth (such as C-section birthing) causing changes in the microbiome, increasing weight gain, and inhibiting intestinal expression of immune genes in neonates. Furthermore, excess antibiotic exposure is associated with the development of neurological and psychiatric disorders. Given the tendency of early perturbations to increase disease risks, it is important to evaluate effects of significant perturbations to microbiome at early ages, such as through antibiotic use.

Currently, no strategies exist to restore the microbiome other than reliance on spontaneous repair mechanism, which often takes months in a healthy individual barring further antibiotic exposure. Modern lifestyle and urban environments, however, work against this spontaneous repair, significantly reducing the microbiome diversity not only generationally but within an individual's lifespan. Contrary to popular belief, ingestion of probiotics, particularly after antibiotics, has been demonstrated to slow down the repair as it introduces an exogenous and massive amounts of only a few types of bacterial strains into a finely-tuned ecosystem of hundreds of different strains.

It is hypothesized that by preserving the child's microbiome prior to antibiotic therapy and reintroducing it afterwards through an autologous fecal matter transplant (FMT) will assist in a quick, effective, and host-specific microbiome recolonization to the levels and patterns to those prior to antibiotics. This would in turn reduce the overall loss of microbiome diversity over the child's lifespan, essentially providing a 'reset' option to the child's most unadulterated version of microbiome.

FMTs have been utilized, including in pediatric populations, to successfully treat recurring Clostridium difficile infections and are being investigated further as an adjunctive treatment in the management of ulcerative colitis, Crohn's Disease, and autism symptoms. Administration of heterologous FMTs (where recipient is different from donor), however, carry their own complexities - stool samples supplied by donors have to be identified and screened and are traditionally delivered in a medical setting as an out-patient procedure. The heterologous FMTs performed today layer the process with additional steps of ideal donor identification and sample screening for possible transmissible pathogens. This proposal uses an autologous sample, which means the sample comes from the healthy child and is administered to the same child after infection and the antibiotic course, conserving the absolutely unique diversity and heritage that that particular child's microbiome had before perturbation due to disease and antibiotics.

In adults, an FMT in form of a capsule for oral use has demonstrated equally successful treatment of C. difficile infection as a rectally-delivered sample. In children, since they cannot swallow capsules, FMTs are delivered as enemas and colonoscopies or through nasogastric and nasojejunal tubes, which require significant resources for the administration of the procedure including anesthesia and observation in addition to the very likely stress impact on the patient.

To evade the invasive nature of these deliveries, novel systems through oral consumption have been investigated. In C-section born infants, maternal stool sample mixed in a bottle of milk and drank by the newborns restored normal gut microbial development to resemble that of vaginally-born babies. The approach utilizes delivering the sample by mixing it in maternal milk or formula and feeding it to the child through a bottle, which can be performed anywhere without any discomfort for the child.

Early life microbiome preservation and restoration holds a tremendous therapeutic potential. Similar to the idea of umbilical stem cells harvesting where stem cells are collected from the infant's umbilical cord, stored, and used as autologous therapeutic transplants in certain cases of cancer, preserved early-life microbiome could be used after antibiotic therapy to restore the composition of the microbiome to the pre-antibiotic state. Unlike the umbilical stem cells harvesting however, fecal sample collection and administration is considerably easier, and the predicted chances for the need of restorative therapy almost certain. Clinical success of such microbiome restorative therapy would exponentially decrease the loss of microbiome diversity and dynamics over one's lifetime, and, by extension, decrease aforementioned associated risks.

The study will be a correlational, case-control study comparing the effects of autologous fecal matter transplant (aFMT) after antibiotic therapy on infant microbiome. The recruitment will be of infants and toddlers up to 4 years of age and of caregivers to collect and freeze fecal samples once a month throughout the duration of the study. The caregivers will be asked to notify the study team if the child has been administered antibiotics, and, after the therapy has ended, the last collected sample prior to treatment will be used for autologous transplant by mixing the frozen infant fecal pellet in milk and administering it to the child. The diversity and composition of the child's fecal microbiome prior and after the transplant will be compared, and then compare those results with the microbiome of control group of children who have received antibiotics but no intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy infants and toddlers 1 month to 4 years of age (regardless of birth mode, sex, or diet (breastmilk, formula, solids, etc.)

Exclusion Criteria:

* Child's antibiotic use within 3 months before inclusion in the study
* Documented immunological condition from the child's pediatrician

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
safety of the autologous FMT measured via questionnaires and medical evaluations | 6 months
  Endpoints: Safety, defined as no/minimal serious adverse effects

SECONDARY OUTCOMES:
microbiome structure during development measured via DNA sequencing | 6 months
  microbiota structure recovery, antibiotic resistance dynamics

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gloria Dominguez-Bello, PhD, Principal Investigator — Rutgers Department of Biochemistry & Microbiology
Locations (1):
- Rutgers Department of Biochemistry & Microbiology, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will not share personal identifiers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: At the time publication of results, DNA sequences will be published as requested by the Journals, in a sequences database (such as ENA, SRA, GenBank, DDBJ).
Access Criteria: Determined by the biological database of computerized ("digital") nucleic acid sequences.

REFERENCES:
- [Background] Korpela K, Helve O, Kolho KL, Saisto T, Skogberg K, Dikareva E, Stefanovic V, Salonen A, Andersson S, de Vos WM. Maternal Fecal Microbiota Transplantation in Cesarean-Born Infants Rapidly Restores Normal Gut Microbial Development: A Proof-of-Concept Study. Cell. 2020 Oct 15;183(2):324-334.e5. doi: 10.1016/j.cell.2020.08.047. Epub 2020 Oct 1. PMID 33007265
- [Background] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074
- [Background] Wang WL, Xu SY, Ren ZG, Tao L, Jiang JW, Zheng SS. Application of metagenomics in the human gut microbiome. World J Gastroenterol. 2015 Jan 21;21(3):803-14. doi: 10.3748/wjg.v21.i3.803. PMID 25624713
- [Background] Kronman MP, Nielson HJ, Adler AL, Giefer MJ, Wahbeh G, Singh N, Zerr DM, Suskind DL. Fecal microbiota transplantation via nasogastric tube for recurrent clostridium difficile infection in pediatric patients. J Pediatr Gastroenterol Nutr. 2015 Jan;60(1):23-6. doi: 10.1097/MPG.0000000000000545. PMID 25162365
- [Background] Martinez KB, Leone V, Chang EB. Western diets, gut dysbiosis, and metabolic diseases: Are they linked? Gut Microbes. 2017 Mar 4;8(2):130-142. doi: 10.1080/19490976.2016.1270811. Epub 2017 Jan 6. PMID 28059614
- [Background] Kang DW, Adams JB, Coleman DM, Pollard EL, Maldonado J, McDonough-Means S, Caporaso JG, Krajmalnik-Brown R. Long-term benefit of Microbiota Transfer Therapy on autism symptoms and gut microbiota. Sci Rep. 2019 Apr 9;9(1):5821. doi: 10.1038/s41598-019-42183-0. PMID 30967657
- [Background] Kang DW, Adams JB, Gregory AC, Borody T, Chittick L, Fasano A, Khoruts A, Geis E, Maldonado J, McDonough-Means S, Pollard EL, Roux S, Sadowsky MJ, Lipson KS, Sullivan MB, Caporaso JG, Krajmalnik-Brown R. Microbiota Transfer Therapy alters gut ecosystem and improves gastrointestinal and autism symptoms: an open-label study. Microbiome. 2017 Jan 23;5(1):10. doi: 10.1186/s40168-016-0225-7. PMID 28122648
- [Background] Suskind DL, Brittnacher MJ, Wahbeh G, Shaffer ML, Hayden HS, Qin X, Singh N, Damman CJ, Hager KR, Nielson H, Miller SI. Fecal microbial transplant effect on clinical outcomes and fecal microbiome in active Crohn's disease. Inflamm Bowel Dis. 2015 Mar;21(3):556-63. doi: 10.1097/MIB.0000000000000307. PMID 25647155
- [Background] Hourigan SK, Chen LA, Grigoryan Z, Laroche G, Weidner M, Sears CL, Oliva-Hemker M. Microbiome changes associated with sustained eradication of Clostridium difficile after single faecal microbiota transplantation in children with and without inflammatory bowel disease. Aliment Pharmacol Ther. 2015 Sep;42(6):741-52. doi: 10.1111/apt.13326. Epub 2015 Jul 21. PMID 26198180
- [Background] Helaly AMN, El-Attar YA, Khalil M, Ahmed Ghorab DSE, El-Mansoury AM. Antibiotic Abuse Induced Histopathological and Neurobehavioral Disorders in Mice. Curr Drug Saf. 2019;14(3):199-208. doi: 10.2174/1574886314666190612130921. PMID 31195950
- [Background] Bonifacio E, Warncke K, Winkler C, Wallner M, Ziegler AG. Cesarean section and interferon-induced helicase gene polymorphisms combine to increase childhood type 1 diabetes risk. Diabetes. 2011 Dec;60(12):3300-6. doi: 10.2337/db11-0729. PMID 22110093
- [Background] Algert CS, McElduff A, Morris JM, Roberts CL. Perinatal risk factors for early onset of Type 1 diabetes in a 2000-2005 birth cohort. Diabet Med. 2009 Dec;26(12):1193-7. doi: 10.1111/j.1464-5491.2009.02878.x. PMID 20002469
- [Background] Marild K, Stephansson O, Montgomery S, Murray JA, Ludvigsson JF. Pregnancy outcome and risk of celiac disease in offspring: a nationwide case-control study. Gastroenterology. 2012 Jan;142(1):39-45.e3. doi: 10.1053/j.gastro.2011.09.047. Epub 2011 Oct 10. PMID 21995948
- [Background] Decker E, Engelmann G, Findeisen A, Gerner P, Laass M, Ney D, Posovszky C, Hoy L, Hornef MW. Cesarean delivery is associated with celiac disease but not inflammatory bowel disease in children. Pediatrics. 2010 Jun;125(6):e1433-40. doi: 10.1542/peds.2009-2260. Epub 2010 May 17. PMID 20478942
- [Background] Kirjavainen PV, Arvola T, Salminen SJ, Isolauri E. Aberrant composition of gut microbiota of allergic infants: a target of bifidobacterial therapy at weaning? Gut. 2002 Jul;51(1):51-5. doi: 10.1136/gut.51.1.51. PMID 12077091
- [Background] Isolauri E, Salminen S; Nutrition, Allergy, Mucosal Immunology, and Intestinal Microbiota (NAMI) Research Group Report. Probiotics: use in allergic disorders: a Nutrition, Allergy, Mucosal Immunology, and Intestinal Microbiota (NAMI) Research Group Report. J Clin Gastroenterol. 2008 Jul;42 Suppl 2:S91-6. doi: 10.1097/MCG.0b013e3181639a98. PMID 18542035
- [Background] Isolauri E, Kalliomaki M, Laitinen K, Salminen S. Modulation of the maturing gut barrier and microbiota: a novel target in allergic disease. Curr Pharm Des. 2008;14(14):1368-75. doi: 10.2174/138161208784480207. PMID 18537659
- [Background] Huurre A, Laitinen K, Rautava S, Korkeamaki M, Isolauri E. Impact of maternal atopy and probiotic supplementation during pregnancy on infant sensitization: a double-blind placebo-controlled study. Clin Exp Allergy. 2008 Aug;38(8):1342-8. doi: 10.1111/j.1365-2222.2008.03008.x. Epub 2008 May 8. PMID 18477013
- [Background] Roduit C, Scholtens S, de Jongste JC, Wijga AH, Gerritsen J, Postma DS, Brunekreef B, Hoekstra MO, Aalberse R, Smit HA. Asthma at 8 years of age in children born by caesarean section. Thorax. 2009 Feb;64(2):107-13. doi: 10.1136/thx.2008.100875. Epub 2008 Dec 3. PMID 19052046
- [Background] Kero J, Gissler M, Gronlund MM, Kero P, Koskinen P, Hemminki E, Isolauri E. Mode of delivery and asthma -- is there a connection? Pediatr Res. 2002 Jul;52(1):6-11. doi: 10.1203/00006450-200207000-00004. PMID 12084840
- [Background] Ege MJ, Mayer M, Normand AC, Genuneit J, Cookson WO, Braun-Fahrlander C, Heederik D, Piarroux R, von Mutius E; GABRIELA Transregio 22 Study Group. Exposure to environmental microorganisms and childhood asthma. N Engl J Med. 2011 Feb 24;364(8):701-9. doi: 10.1056/NEJMoa1007302. PMID 21345099
- [Background] Couzin-Frankel J. Bacteria and asthma: untangling the links. Science. 2010 Nov 26;330(6008):1168-9. doi: 10.1126/science.330.6008.1168. No abstract available. PMID 21109643
- [Background] Murphy R, Stewart AW, Braithwaite I, Beasley R, Hancox RJ, Mitchell EA; ISAAC Phase Three Study Group. Antibiotic treatment during infancy and increased body mass index in boys: an international cross-sectional study. Int J Obes (Lond). 2014 Aug;38(8):1115-9. doi: 10.1038/ijo.2013.218. Epub 2013 Nov 21. PMID 24257411
- [Background] Trasande L, Blustein J, Liu M, Corwin E, Cox LM, Blaser MJ. Infant antibiotic exposures and early-life body mass. Int J Obes (Lond). 2013 Jan;37(1):16-23. doi: 10.1038/ijo.2012.132. Epub 2012 Aug 21. PMID 22907693
- [Background] Blustein J, Attina T, Liu M, Ryan AM, Cox LM, Blaser MJ, Trasande L. Association of caesarean delivery with child adiposity from age 6 weeks to 15 years. Int J Obes (Lond). 2013 Jul;37(7):900-6. doi: 10.1038/ijo.2013.49. Epub 2013 Apr 8. PMID 23670220
- [Background] Ajslev TA, Andersen CS, Gamborg M, Sorensen TI, Jess T. Childhood overweight after establishment of the gut microbiota: the role of delivery mode, pre-pregnancy weight and early administration of antibiotics. Int J Obes (Lond). 2011 Apr;35(4):522-9. doi: 10.1038/ijo.2011.27. Epub 2011 Mar 8. PMID 21386800
- [Background] Korpela K, Salonen A, Virta LJ, Kekkonen RA, Forslund K, Bork P, de Vos WM. Intestinal microbiome is related to lifetime antibiotic use in Finnish pre-school children. Nat Commun. 2016 Jan 26;7:10410. doi: 10.1038/ncomms10410. PMID 26811868
- [Background] Rogawski ET, Platts-Mills JA, Seidman JC, John S, Mahfuz M, Ulak M, Shrestha SK, Soofi SB, Yori PP, Mduma E, Svensen E, Ahmed T, Lima AA, Bhutta ZA, Kosek MN, Lang DR, Gottlieb M, Zaidi AK, Kang G, Bessong PO, Houpt ER, Guerrant RL. Use of antibiotics in children younger than two years in eight countries: a prospective cohort study. Bull World Health Organ. 2017 Jan 1;95(1):49-61. doi: 10.2471/BLT.16.176123. Epub 2016 Nov 3. PMID 28053364